CLINICAL TRIAL: NCT02953639
Title: A Phase IIb, Multicenter, Randomized, Double-Blind, Parallel Group, Placebo Controlled Study to Evaluate the Efficacy, Safety and Tolerability of Basmisanil (RO5186582) as Adjunctive Treatment in Patients With Cognitive Impairment Associated With Schizophrenia Treated With Antipsychotics
Brief Title: A Study to Evaluate the Effects of Basmisanil in Participants With Cognitive Impairment Associated With Schizophrenia (CIAS) Treated With Antipsychotics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP39207
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — basmisanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received matching Placebo to Basmisanil orally twice daily for 24 weeks.
  Interventions: Drug: Placebo
- Basmisanil 80mg BID (Experimental): Participants received Basmisanil 80 mg orally twice daily (BID) for 24 weeks.
  Interventions: Drug: Basmisanil
- Basmisanil 240mg BID (Experimental): Participants received Basmisanil 240 mg orally twice daily (BID) for 24 weeks.
  Interventions: Drug: Basmisanil

INTERVENTIONS:
Drug: Basmisanil — Participants received either 80 milligrams (mg) or 240 mg of Basmisanil, as per the dosing schedules described above.
  Arms: Basmisanil 240mg BID; Basmisanil 80mg BID
Drug: Placebo — Participants received matching Placebo to Basmisanil, as per the dosing schedules described above.
  Arms: Placebo

SUMMARY:
This multicenter study assessed the effects of 24 weeks of basmisanil treatment on cognition and functioning of stable schizophrenia participants treated with antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia of any type utilizing the Mini International Neuropsychiatric Interview and diagnostic and statistical manual of mental disorders, fifth edition (DSM-5) direct clinical assessments, family informants and past medical records
* Evidence of stability of symptoms for 3 months at screening, that is, without hospitalizations for schizophrenia or increase in level of psychiatric care due to worsening of symptoms of schizophrenia
* Participants with schizophrenia clinical symptom severity defined by the following: hallucinatory behavior item score less than or equal to (</=) 5 and a delusion item score </= 5 of the PANSS
* Participants on a stable regimen of antipsychotic therapy for at least 3 months at screening and receiving no more than two antipsychotics

Exclusion Criteria:

* Participants with current DSM-5 diagnosis other than schizophrenia including bipolar disorder, schizoaffective disorder and major depressive disorder
* Clinically significant neurological illness or significant head trauma that affects cognitive function, in the judgment of the principal investigator
* Full scale intelligence quotient </=65 on the Wechsler Abbreviated Scale of Intelligence at screening
* Positive result at screening for hepatitis B, hepatitis C, or human immunodeficiency virus-1 and 2
* Moderate to severe substance use disorder (other than nicotine or caffeine), as defined by the DSM-5, within the last 12 months
* Suicide attempt within 1 year or currently at risk of suicide in the opinion of the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 214 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- United States (37):
  - Woodland International Research Group Inc., Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - California Clinical Trials, Glendale, California
  - Alliance for Wellness, dba Alliance for Research, Long Beach, California
  - Synergy Clinical Research, National City, California
  - Pacific Research Partners, LLC, Oakland, California
  - NRC Research Institute, Orange, California
  - CNRI - Los Angeles, LLC, Pico Rivera, California
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - Collaborative Neuroscience Network Inc., Torrance, California
  - Yale School of Medicine - CT Mental Health Center (CMHC) - Schizophrenia Research Clinic, New Haven, Connecticut
  - Vantage Clinical Trials, Largo, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Meridien Research, Maitland, Florida
  - University of Miami Dept of Psychiatry, Miami, Florida
  - Behavioral Clinical Research, Inc., North Miami, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Booker, J. Gary, MD, APMC, Shreveport, Louisiana
  - Louisiana Clinical Research, LLC, Shreveport, Louisiana
  - CBH Health, Gaithersburg, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Arch Clinical Trials, LLC, St Louis, Missouri
  - St Louis Clinical Trials, St Louis, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Manhattan Psychiatric Center; Psychopharmacology Research Unit, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - University Hospitals, Cleveland, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Pillar Clinical Research LLC, Garland, Texas
  - University Hills Clinical Research - Irving;Office of Dr. Knesevich, Irving, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 37 centers in 1 country.
Pre-assignment Details: Overall, 214 participants were enrolled into the study across 37 sites in the US. Of these, 213 participants received study treatment and were included in the Intent-To-Treat (ITT) and Safety populations. One participant randomized to the placebo arm withdrew prior to the first study treatment administration.
Period: Overall Study
Arm/Group | Placebo | Basmisanil 80mg BID | Basmisanil 240mg BID
Started | 81 | 54 | 78
Completed | 61 | 40 | 62
Not Completed | 20 | 14 | 16
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Lost to Follow-up | 8 | 4 | 3
Not completed — Non-Compliance With Study Drug | 0 | 2 | 1
Not completed — Multiple Reasons | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 8 | 10
Not completed — Completed or Discontinued information is missing | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Basmisanil 80mg BID | Basmisanil 240mg BID | Total
Number analyzed (Participants) | 81 | 54 | 78 | 213
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.4 (8.2) | 36.8 (8.6) | 37.4 (8.4) | 36.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 18 | 50
  Male | 61 | 42 | 60 | 163
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 13 | 7 | 12 | 32
  Not Hispanic or Latino | 68 | 47 | 66 | 181
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 3 | 0 | 2 | 5
  Black or African American | 51 | 30 | 51 | 132
  MULTIPLE | 1 | 0 | 0 | 1
  UNKNOWN | 1 | 1 | 2 | 4
  White | 25 | 23 | 23 | 71

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in MATRICS Consensus Cognitive Battery (MCCB) Neurocognitive Composite Score
Description: The MCCB is a cognitive battery to assess 7 domains recommended by the MATRICS initiative (i.e., working memory, verbal learning, speed of processing, attention/vigilance, visual learning, social cognition, reasoning and problem solving). The MCCB neurocognitive composite T-score is a standardized mean of the six domain scores (excluding social cognition). Raw scores are converted to age and sex adjusted t-scores which are standardized to normative data, and have a mean of 50 and standard deviation of 10 in the general healthy population. A higher composite T-score represents lower impairment.
Time Frame: Baseline up to Week 24
Population: The EAP2 Population was defined as all participants in the Efficacy Analysis Population (EAP) who were randomized to placebo or 240mg Basmisanil (excluded participants randomized to 80mg Basmisanil due to the results of a futility analysis which meant that enrolment into the 80mg Basmisanil arm was discontinued). Data presented below is only for participants that were included in the actual analysis.
Measure: Mean (Standard Deviation); unit: Composite T-Score
Arm/Group | Placebo | Basmisanil 240mg BID
Number analyzed (Participants) | 76 | 77
Composite T-Score
  Baseline | 32.50 (14.47) | 32.36 (11.44)
  Week 12 Day 84: number analyzed (Participants) | 58 | 58
  Week 12 Day 84 | -0.17 (5.07) | -0.28 (6.08)
  Week 24 Day 168: number analyzed (Participants) | 52 | 45
  Week 24 Day 168 | 1.08 (5.78) | 1.36 (4.80)
Statistical Analysis 1: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84; Test type: Superiority; p = 0.730, Mixed Models Analysis; Treatment Difference = -0.36, 90% CI 2-sided [-2.11 to 1.38]
Statistical Analysis 2: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168; Test type: Superiority; p = 0.793, Mixed Models Analysis; Treatment Difference = 0.28, 90% CI 2-sided [-1.47 to 2.02]

2. Secondary Outcome: Change From Baseline to Week 24 in MCCB Cognitive Domain Scores
Description: The MCCB is a cognitive battery to assess 7 domains recommended by the MATRICS initiative (i.e., working memory, verbal learning, speed of processing, attention/vigilance, visual learning, social cognition, reasoning and problem solving). Raw scores are converted to age and sex adjusted t-scores which are standardized to normative data, and have a mean of 50 and standard deviation of 10 in the general healthy population. A higher T-score represents lower impairment.
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Basmisanil 240mg BID
Number analyzed (Participants) | 76 | 77
T-score
  Baseline (Attention/Vigilance) | 40.75 (12.31) | 39.66 (12.08)
  Week 12 Day 84 (Attention/Vigilance): number analyzed (Participants) | 58 | 58
  Week 12 Day 84 (Attention/Vigilance) | -0.16 (8.00) | -0.14 (8.80)
  Week 24 Day 168 (Attention/Vigilance): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (Attention/Vigilance) | 0.63 (6.89) | 0.51 (8.49)
  Baseline (Reasoning and Problem Solving) | 42.75 (12.61) | 43.71 (10.12)
  Week 12 Day 84 (Reasoning and Problem Solving): number analyzed (Participants) | 58 | 58
  Week 12 Day 84 (Reasoning and Problem Solving) | 0.05 (8.94) | 0.05 (6.07)
  Week 24 Day 168 (Reasoning and Problem Solving): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (Reasoning and Problem Solving) | 1.69 (7.23) | 2.18 (6.13)
  Baseline (Social Cognition) | 37.79 (13.30) | 38.38 (13.09)
  Week 12 Day 84 (Social Cognition): number analyzed (Participants) | 58 | 58
  Week 12 Day 84 (Social Cognition) | 0.62 (7.74) | -0.62 (8.55)
  Week 24 Day 168 (Social Cognition): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (Social Cognition) | -1.71 (7.24) | 0.96 (7.10)
  Baseline (Speed of Processing) | 37.08 (13.10) | 37.81 (12.70)
  Week 12 Day 84 (Speed of Processing): number analyzed (Participants) | 58 | 58
  Week 12 Day 84 (Speed of Processing) | -1.48 (7.41) | -1.66 (6.07)
  Week 24 Day 168 (Speed of Processing): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (Speed of Processing) | 0.37 (6.85) | 0.13 (4.88)
  Baseline (Verbal Learning) | 37.34 (9.20) | 36.53 (7.41)
  Week 12 Day 84 (Verbal Learning): number analyzed (Participants) | 58 | 58
  Week 12 Day 84 (Verbal Learning) | 0.26 (7.99) | 0.45 (7.01)
  Week 24 Day 168 (Verbal Learning): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (Verbal Learning) | 0.46 (8.33) | 0.36 (6.53)
  Baseline (Visual Learning) | 35.96 (12.18) | 35.38 (11.98)
  Week 12 Day 84 (Visual Learning): number analyzed (Participants) | 58 | 58
  Week 12 Day 84 (Visual Learning) | -0.91 (8.14) | -0.48 (9.35)
  Week 24 Day 168 (Visual Learning): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (Visual Learning) | -0.98 (8.56) | 0.53 (9.33)
  Baseline (Working Memory) | 35.99 (12.56) | 36.23 (10.09)
  Week 12 Day 84 (Working Memory): number analyzed (Participants) | 58 | 58
  Week 12 Day 84 (Working Memory) | 1.62 (6.99) | 0.76 (6.41)
  Week 24 Day 168 (Working Memory): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (Working Memory) | 2.37 (6.34) | 1.76 (6.68)
Statistical Analysis 1: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (Attention/Vigilance); Test type: Superiority; p = 0.556, Mixed Models Analysis; Treatment Difference = -0.91, 90% CI 2-sided [-3.46 to 1.64]
Statistical Analysis 2: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (Attention/Vigilance); Test type: Superiority; p = 0.848, Mixed Models Analysis; Treatment Difference = -0.27, 90% CI 2-sided [-2.59 to 2.05]
Statistical Analysis 3: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (Reasoning and Problem Solving); Test type: Superiority; p = 0.973, Mixed Models Analysis; Treatment Difference = 0.04, 90% CI 2-sided [-2.08 to 2.16]
Statistical Analysis 4: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (Reasoning and Problem Solving); Test type: Superiority; p = 0.651, Mixed Models Analysis; Treatment Difference = 0.57, 90% CI 2-sided [-1.53 to 2.67]
Statistical Analysis 5: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (Social Cognition); Test type: Superiority; p = 0.350, Mixed Models Analysis; Treatment Difference = -1.44, 90% CI 2-sided [-3.89 to 1.08]
Statistical Analysis 6: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (Social Cognition); Test type: Superiority; p = 0.121, Mixed Models Analysis; Treatment Difference = 2.18, 90% CI 2-sided [-0.14 to 4.50]
Statistical Analysis 7: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (Speed of Processing); Test type: Superiority; p = 0.911, Mixed Models Analysis; Treatment Difference = -0.13, 90% CI 2-sided [-2.10 to 1.83]
Statistical Analysis 8: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (Speed of Processing); Test type: Superiority; p = 0.987, Mixed Models Analysis; Treatment Difference = 0.02, 90% CI 2-sided [-1.99 to 2.03]
Statistical Analysis 9: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (Verbal Learning); Test type: Superiority; p = 0.803, Mixed Models Analysis; Treatment Difference = -0.34, 90% CI 2-sided [-2.62 to 1.93]
Statistical Analysis 10: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (Verbal Learning); Test type: Superiority; p = 0.502, Mixed Models Analysis; Treatment Difference = -0.94, 90% CI 2-sided [-3.26 to 1.38]
Statistical Analysis 11: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (Visual Learning); Test type: Superiority; p = 0.945, Mixed Models Analysis; Treatment Difference = -0.11, 90% CI 2-sided [-2.74 to 2.52]
Statistical Analysis 12: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (Visual Learning); Test type: Superiority; p = 0.488, Mixed Models Analysis; Treatment Difference = 1.11, 90% CI 2-sided [-1.54 to 3.76]
Statistical Analysis 13: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (Working Memory); Test type: Superiority; p = 0.262, Mixed Models Analysis; Treatment Difference = -1.37, 90% CI 2-sided [-3.38 to 0.64]
Statistical Analysis 14: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (Working Memory); Test type: Superiority; p = 0.489, Mixed Models Analysis; Treatment Difference = -0.89, 90% CI 2-sided [-3.01 to 1.23]

3. Secondary Outcome: Change From Baseline to Week 24 in Wechsler Memory Scale Fourth Edition, Verbal Paired Associates (WMS IV-PAL) Score
Description: The Paired Associates Learning (PAL I and II) of the WMS-IV (Wechsler Memory Scale Fourth edition) is a test of verbal learning and memory that requires the participant to learn novel word pairs. The participant learns the word pairs across learning trials and is asked to recall them immediately (PAL I) or after a 30-minute delay (PAL II). Data is presented here for 3 Scores: VPA I total raw score, VPA II total raw score and VPA II Recognition total raw score. The total raw score ranges for these 3 Scores are 0 to 56, 0 to 14 and 0 to 40 respectively, with larger total raw scores indicating better performance.
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Basmisanil 240mg BID
Number analyzed (Participants) | 76 | 77
Scores on a Scale
  Baseline (VPA I total raw score) | 31.14 (12.53) | 32.30 (11.75)
  Week 12 Day 84 (VPA I total raw score): number analyzed (Participants) | 58 | 58
  Week 12 Day 84 (VPA I total raw score) | 2.14 (6.55) | 0.36 (7.33)
  Week 24 Day 168 (VPA I total raw score): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (VPA I total raw score) | 4.42 (6.58) | 5.09 (6.40)
  Baseline (VPA II total raw score) | 9.25 (3.76) | 9.77 (3.54)
  Week 12 Day 84 (VPA II total raw score): number analyzed (Participants) | 58 | 58
  Week 12 Day 84 (VPA II total raw score) | 0.12 (2.29) | 0.26 (2.15)
  Week 24 Day 168 (VPA II total raw score): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (VPA II total raw score) | 0.69 (2.16) | 1.60 (2.33)
  Baseline (VPA II recognition total raw score): number analyzed (Participants) | 75 | 76
  Baseline (VPA II recognition total raw score) | 36.24 (5.37) | 37.36 (5.12)
  Week 12 Day 84 (VPA II recognition total raw score): number analyzed (Participants) | 56 | 58
  Week 12 Day 84 (VPA II recognition total raw score) | 0.48 (5.43) | -0.55 (2.92)
  Week 24 Day 168 (VPA II recognition total raw score): number analyzed (Participants) | 50 | 44
  Week 24 Day 168 (VPA II recognition total raw score) | 1.12 (5.60) | 0.36 (2.80)
Statistical Analysis 1: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (VPA I total raw score); Test type: Superiority; p = 0.211, Mixed Models Analysis; Treatment Difference = -1.63, 90% CI 2-sided [-3.78 to 0.52]
Statistical Analysis 2: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (VPA I total raw score); Test type: Superiority; p = 0.787, Mixed Models Analysis; Treatment Difference = 0.35, 90% CI 2-sided [-1.81 to 2.52]
Statistical Analysis 3: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (VPA II total raw score); Test type: Superiority; p = 0.477, Mixed Models Analysis; Treatment Difference = 0.28, 90% CI 2-sided [-0.37 to 0.94]
Statistical Analysis 4: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (VPA II total raw score); Test type: Superiority; p = 0.028, Mixed Models Analysis; Treatment Difference = 0.91, 90% CI 2-sided [0.23 to 1.58]
Statistical Analysis 5: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (VPA II recognition total raw score); Test type: Superiority; p = 0.683, Mixed Models Analysis; Treatment Difference = -0.30, 90% CI 2-sided [-1.51 to 0.91]
Statistical Analysis 6: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (VPA II recognition total raw score); Test type: Superiority; p = 0.954, Mixed Models Analysis; Treatment Difference = 0.04, 90% CI 2-sided [-1.13 to 1.22]

4. Secondary Outcome: Change From Baseline to Week 24 in Wechsler Memory Scale Fourth Edition, Logical Memory Test (WMS IV-LM) Score
Description: Logical memory (LM) assesses narrative memory under free-recall conditions. Two short stories are presented orally. The examinee is asked to retell each story from memory immediately after hearing it (LM I). In the delayed condition (LM II), the examinee is asked to retell both stories from the immediate condition (delayed free recall). Data is presented here for 2 Scores: LM I total raw score and LM II total raw score. The total raw score range is from 0 to 50 with larger total raw scores indicating better performance.
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Basmisanil 240mg BID
Number analyzed (Participants) | 76 | 77
Scores on a Scale
  Baseline (LM I) | 16.55 (5.80) | 16.22 (8.13)
  Week 12 Day 84 (LM I): number analyzed (Participants) | 58 | 58
  Week 12 Day 84 (LM I) | -2.60 (5.33) | -0.83 (5.66)
  Week 24 Day 168 (LM I): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (LM I) | -3.02 (4.96) | -2.29 (5.29)
  Baseline (LM II) | 13.72 (6.57) | 14.29 (8.22)
  Week 12 Day 84 (LM II): number analyzed (Participants) | 58 | 56
  Week 12 Day 84 (LM II) | -2.91 (6.04) | -2.63 (6.08)
  Week 24 Day 168 (LM II): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (LM II) | -2.73 (4.94) | -3.22 (5.15)
Statistical Analysis 1: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (LM I); Test type: Superiority; p = 0.164, Mixed Models Analysis; Treatment Difference = 1.45, 90% CI 2-sided [-0.27 to 3.17]
Statistical Analysis 2: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (LM I); Test type: Superiority; p = 0.559, Mixed Models Analysis; Treatment Difference = 0.56, 90% CI 2-sided [-1.02 to 2.14]
Statistical Analysis 3: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (LM II); Test type: Superiority; p = 0.912, Mixed Models Analysis; Treatment Difference = 0.12, 90% CI 2-sided [-1.70 to 1.94]
Statistical Analysis 4: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (LM II); Test type: Superiority; p = 0.706, Mixed Models Analysis; Treatment Difference = -0.36, 90% CI 2-sided [-1.93 to 1.22]

5. Secondary Outcome: Change From Baseline to Week 24 in Ratio Between Trail Making Test (TMT)- Part B and TMT- Part A Scores
Description: The TMT consists of two parts: Trail Making Part A, which is a part of the standard MCCB and Trail Making Part B additionally included in this study. Circles containing numbers (Part A) or both numbers and letters (Part B) must be sequentially connected. The difference (ratio) in performance between Part A and Part B reflects executive processes and will be used to assess executive functioning including cognitive set shifting abilities and data for this ratio is presented here. Smaller ratio values, hence decreases from baseline (TMT-B/TMT-A ratio values below 1) indicate higher executive functioning capabilities.
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | Basmisanil 240mg BID
Number analyzed (Participants) | 76 | 77
Ratio
  Baseline | 3.27 (1.65) | 3.12 (1.58)
  Week 12 Day 84: number analyzed (Participants) | 56 | 56
  Week 12 Day 84 | -0.37 (1.19) | -0.12 (1.34)
  Week 24 Day 168: number analyzed (Participants) | 50 | 43
  Week 24 Day 168 | -0.23 (2.00) | -0.06 (1.22)
Statistical Analysis 1: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84; Test type: Superiority; p = 0.527, Mixed Models Analysis; Treatment Difference = 1.04, 90% CI 2-sided [0.94 to 1.15]
Statistical Analysis 2: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168; Test type: Superiority; p = 0.636, Mixed Models Analysis; Treatment Difference = 1.04, 90% CI 2-sided [0.92 to 1.17]

6. Secondary Outcome: Change From Baseline to Week 24 in Personal and Social Performance (PSP) Total Score
Description: The PSP Total Score is an integer result in the range of 0 to 100. Larger values, hence increases from baseline in the PSP total score, indicate higher social and personal functioning.
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Basmisanil 240mg BID
Number analyzed (Participants) | 74 | 76
Scores on a Scale
  Baseline | 59.82 (11.88) | 60.88 (10.87)
  Week 12 Day 84: number analyzed (Participants) | 55 | 57
  Week 12 Day 84 | 3.13 (8.30) | 2.26 (8.68)
  Week 24 Day 168: number analyzed (Participants) | 51 | 44
  Week 24 Day 168 | 3.75 (9.66) | 4.14 (10.05)
Statistical Analysis 1: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84; Test type: Superiority; p = 0.323, Mixed Models Analysis; Treatment Difference = -1.36, 90% CI 2-sided [-3.63 to 0.91]
Statistical Analysis 2: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168; Test type: Superiority; p = 0.579, Mixed Models Analysis; Treatment Difference = -0.95, 90% CI 2-sided [-3.77 to 1.88]

7. Secondary Outcome: Change From Baseline to Week 24 in Schizophrenia Cognition Rating Scale (SCoRS) Total Score
Description: The main parameter of interest for the Schizophrenia Cognition Rating Scale (SCoRS) is the SCoRS 'Total Score'. The total score range is from 0 to 80 with lower scores indicating better day-to-day functioning.
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Basmisanil 240mg BID
Number analyzed (Participants) | 76 | 77
Scores on a Scale
  Baseline | 37.07 (8.52) | 36.53 (9.84)
  Week 12 Day 84: number analyzed (Participants) | 58 | 58
  Week 12 Day 84 | -2.91 (6.06) | -3.66 (5.78)
  Week 24 Day 168: number analyzed (Participants) | 51 | 45
  Week 24 Day 168 | -3.71 (7.19) | -4.02 (7.79)
Statistical Analysis 1: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84; Test type: Superiority; p = 0.493, Mixed Models Analysis; Treatment Difference = -0.67, 90% CI 2-sided [-2.27 to 0.94]
Statistical Analysis 2: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168; Test type: Superiority; p = 0.926, Mixed Models Analysis; Treatment Difference = -0.12, 90% CI 2-sided [-2.32 to 2.07]

8. Secondary Outcome: Change From Baseline to Week 24 in Clinical Global Impression Severity (CGI-S) Rating
Description: Values for the CGI-S Scale are encoded by the numerical values from 1 to 7 respectively. Higher numerical values represent greater impairment.
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Basmisanil 240mg BID
Number analyzed (Participants) | 75 | 77
Scores on a Scale
  Baseline | 2.45 (0.62) | 2.39 (0.75)
  Week 12 Day 84: number analyzed (Participants) | 57 | 58
  Week 12 Day 84 | -0.21 (0.67) | -0.24 (0.60)
  Week 24 Day 168: number analyzed (Participants) | 52 | 45
  Week 24 Day 168 | -0.19 (0.56) | -0.29 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84; Test type: Superiority; p = 0.839, Mixed Models Analysis; Treatment Difference = -0.02, 90% CI 2-sided [-0.22 to 0.17]
Statistical Analysis 2: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168; Test type: Superiority; p = 0.625, Mixed Models Analysis; Treatment Difference = -0.06, 90% CI 2-sided [-0.27 to 0.15]

9. Secondary Outcome: Change From Baseline to Week 24 in Clinical Global Impression Improvement (CGI-I) Rating
Description: Values for the CGI-I Scale are encoded by the numerical values from 1 to 7 respectively. Higher numerical values represent greater impairment.
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Basmisanil 240mg BID
Number analyzed (Participants) | 58 | 58
Scores on a Scale
  Week 12 Day 84 | -0.45 (0.86) | -0.45 (0.86)
  Week 24 Day 168: number analyzed (Participants) | 52 | 45
  Week 24 Day 168 | -0.62 (1.01) | -0.64 (0.91)
Statistical Analysis 1: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84; Test type: Superiority; p = 0.865, Mixed Models Analysis; Treatment Difference = -0.03, 90% CI 2-sided [-0.28 to 0.23]
Statistical Analysis 2: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168; Test type: Superiority; p = 0.964, Mixed Models Analysis; Treatment Difference = -0.01, 90% CI 2-sided [-0.31 to 0.29]

10. Secondary Outcome: Change From Baseline to Week 24 in Schizophrenia Quality of Life Scale (SQLS)
Description: The SQLS is a patient reported scale consisting of 33 items: 2 domain scores (Cognition & Vitality Score [SQLS-CV] and Psycho-social Score [SQLS-P]) as well as a Total score (SQLS-T) are derived. The overall score range is from 0 to 100. On all scales, higher scores represent a lower quality of life.
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Basmisanil 240mg BID
Number analyzed (Participants) | 76 | 77
Scores on a Scale
  Baseline (SQLS Cognition & Vitality Score): number analyzed (Participants) | 76 | 76
  Baseline (SQLS Cognition & Vitality Score) | 33.81 (17.41) | 34.21 (18.59)
  Week 12 Day 84 (SQLS Cognition & Vitality Score): number analyzed (Participants) | 57 | 58
  Week 12 Day 84 (SQLS Cognition & Vitality Score) | -2.26 (12.66) | 0.21 (14.00)
  Week 24 Day 168 (SQLS Cognition & Vitality Score): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (SQLS Cognition & Vitality Score) | -0.78 (15.71) | -4.32 (13.59)
  Baseline (SQLS Psychosocial Score) | 31.48 (20.26) | 30.84 (20.88)
  Week 12 Day 84 (SQLS Psychosocial Score): number analyzed (Participants) | 57 | 58
  Week 12 Day 84 (SQLS Psychosocial Score) | -0.88 (12.42) | 0.80 (14.49)
  Week 24 Day 168 (SQLS Psychosocial Score): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (SQLS Psychosocial Score) | -1.78 (12.87) | -1.58 (13.27)
  Baseline (SQLS Total Score): number analyzed (Participants) | 76 | 76
  Baseline (SQLS Total Score) | 32.40 (18.51) | 32.14 (19.19)
  Week 12 Day 84 (SQLS Total Score): number analyzed (Participants) | 57 | 58
  Week 12 Day 84 (SQLS Total Score) | -1.42 (11.80) | 0.57 (12.98)
  Week 24 Day 168 (SQLS Total Score): number analyzed (Participants) | 52 | 45
  Week 24 Day 168 (SQLS Total Score) | -1.38 (12.89) | -2.66 (12.31)
Statistical Analysis 1: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (SQLS Cognition & Vitality Score); Test type: Superiority; p = 0.142, Mixed Models Analysis; Treatment Difference = 3.27, 90% CI 2-sided [-0.40 to 6.95]
Statistical Analysis 2: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (SQLS Cognition & Vitality Score); Test type: Superiority; p = 0.416, Mixed Models Analysis; Treatment Difference = -2.32, 90% CI 2-sided [-7.04 to 2.40]
Statistical Analysis 3: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (SQLS Psychosocial Score); Test type: Superiority; p = 0.394, Mixed Models Analysis; Treatment Difference = 1.98, 90% CI 2-sided [-1.86 to 5.83]
Statistical Analysis 4: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (SQLS Psychosocial Score); Test type: Superiority; p = 0.776, Mixed Models Analysis; Treatment Difference = 0.71, 90% CI 2-sided [-3.44 to 4.87]
Statistical Analysis 5: Comparison: Placebo vs Basmisanil 240mg BID; Week 12 Day 84 (SQLS Total Score); Test type: Superiority; p = 0.254, Mixed Models Analysis; Treatment Difference = 2.43, 90% CI 2-sided [-1.09 to 5.94]
Statistical Analysis 6: Comparison: Placebo vs Basmisanil 240mg BID; Week 24 Day 168 (SQLS Total Score); Test type: Superiority; p = 0.816, Mixed Models Analysis; Treatment Difference = -0.57, 90% CI 2-sided [-4.64 to 3.50]

11. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events.
Time Frame: Baseline up to 4 weeks after the last dose of study drug (up to 28 weeks)
Population: The Safety-evaluable population was defined as all participants who received at least one dose of study medication, whether prematurely withdrawn from the study or not. Data are summarized according to actual treatment arm participants were randomized to.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Basmisanil 80mg BID | Basmisanil 240mg BID
Number analyzed (Participants) | 81 | 54 | 78
Percentage of Participants | 39.5 | 46.3 | 48.7

12. Secondary Outcome: Apparent Clearance of Basmisanil at Steady State (CL/F,ss)
Description: Population PK model estimated apparent oral clearance of Basmisanil at steady-state.
Time Frame: Pre-dose (hour 0) in Days 7, 14, 42, 84, 168
Population: Please note that for this Outcome Measure, incomplete PK data was collected as a result of early termination of the study which meant that data for the (CL/F,ss) parameter could not be generated via the Population PK model.
Arm/Group | Basmisanil 80mg BID | Basmisanil 240mg BID
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Apparent Volume of Distribution of Basmisanil at Steady State (Vz/F,ss)
Description: Population PK model estimated apparent volume of distribution of Basmisanil at steady-state.
Time Frame: Pre-dose (hour 0) in Days 7, 14, 42, 84, 168
Population: Please note that for this Outcome Measure, incomplete PK data was collected as a result of early termination of the study which meant that data for the (Vz/F,ss) parameter could not be generated via the Population PK model.
Arm/Group | Basmisanil 80mg BID | Basmisanil 240mg BID
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Area Under the Curve of Basmisanil at Steady State (AUC,ss)
Description: Population PK model estimated AUC of Basmisanil at steady-state.
Time Frame: Pre-dose (hour 0) in Days 7, 14, 42, 84, 168
Population: The Safety-evaluable population was defined as all participants who received at least one dose of study medication, whether prematurely withdrawn from the study or not. Data are summarized according to actual treatment arm participants were randomized to. Data presented below is only for participants included in the actual analysis.
Measure: Median (Full Range); unit: ng*mL/hr
Arm/Group | Basmisanil 80mg BID | Basmisanil 240mg BID
Number analyzed (Participants) | 54 | 78
ng*mL/hr | 41640 [31464 to 51816] | 87624 [66504 to 108768]

15. Secondary Outcome: Maximum Plasma Concentration of Basmisanil at Steady State (Cmax,ss)
Description: Population PK model estimated maximum plasma concentration of Basmisanil at steady-state (ss).
Time Frame: Pre-dose (hour 0) in Days 7, 14, 42, 84, 168
Population: as for outcome 14
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Basmisanil 80mg BID | Basmisanil 240mg BID
Number analyzed (Participants) | 54 | 78
ng/mL | 2079 [1645 to 2513] | 4374 [3455 to 5294]

ADVERSE EVENTS:
Time Frame: Baseline up to 4 weeks after the last dose of study drug (up to 28 weeks)
Arm/Group | Placebo | Basmisanil 80mg BID | Basmisanil 240mg BID
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/54 | 0/78
Serious Adverse Events (participants affected / at risk) | 5/81 | 0/54 | 4/78
Other Adverse Events (participants affected / at risk) | 10/81 | 10/54 | 12/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Basmisanil 80mg BID (N=54) | Basmisanil 240mg BID (N=78)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (2) | 0 (0) | 2 (2)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Basmisanil 80mg BID (N=54) | Basmisanil 240mg BID (N=78)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (4) | 2 (2)
Fatigue (General disorders) | 6 (7) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 7 (9)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)

LIMITATIONS AND CAVEATS:
Following a planned futility analysis, enrolment into the 80mg Basmisanil arm was discontinued as of 8th November 2018. Results from the 80mg Basmisanil arm are thus not presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT02953639/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT02953639/SAP_001.pdf